CLINICAL TRIAL: NCT04994561
Title: Pilot Study to Test the Safety and Efficacy of Metformin, Dasatinib, Rapamycin and Nutritional Supplements (Bio-quercetin; Bio-fisetin; Glucosamine; Nicotinamide Riboside; Trans-resveratrol) in Reducing Clinical Measures of Aging in Older Adults
Brief Title: VIAging Deceleration Trial Using Metformin, Dasatinib, Rapamycin and Nutritional Supplements
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Study was withdrawn
Sponsor: Vitality in Aging Research Group, Inc. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VIA-004
Record Dates: First submitted 2021-07-23; First posted 2021-08-06 (Actual); Last update posted 2022-06-07 (Actual); Status verified 2022-06

CONDITIONS: Aging
Keywords: Aging; Cell senescence
MeSH Terms: interventions — Dietary Supplements; Metformin; Dasatinib; Sirolimus; Glucosamine; nicotinamide-beta-riboside; Resveratrol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Subjects receiving study drugs and nutritional supplements (Experimental): All eligible and consented subjects will receive study drugs and nutritional supplements as described in the intervention.
  Interventions: Drug: Study Drugs and Nutritional Supplements

INTERVENTIONS:
Drug: Study Drugs and Nutritional Supplements — Step 1: 500 mg of metformin and increase their dose 500 mg every 2 weeks up to 2000 mg or until tolerable.
  Step 2: Once at tolerable daily metformin dose, subjects will take 140 mg of dasatinib along with 58 mg to 174 mg (based on body weight) bio-quercetin and 44.5 mg bio-fisetin. Subjects will take dasatinib, bio-quercetin and bio-fisetin for 2 consecutive days as described 4 times over one year (every 3 months) while participating on this study.
  Step 3: Two weeks after the first dasatinib dose is complete, subjects will start taking daily nutritional supplements of 1,500 mg glucosamine, 600 mg nicotinamide riboside and 500 mg trans-resveratrol.
  Step 4: Two weeks after starting daily supplements in Step 3, subjects will take a once weekly 6 mg dose of rapamycin.
  Once subject is taking rapamycin, they will continue on this intervention for 12 months.
  Other Names: metformin, dasatinib, rapamycin and nutritional supplements (bio-quercetin; bio-fisetin; glucosamine; nicotinamide riboside; trans-resveratrol)

SUMMARY:
This study aims to assess the safety and efficacy of study drugs and supplements on clinical (structural and functional) signs of aging and to explore/identify other possible biological measures of aging.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects 65 years of age or older
2. Received full dose of COVID-19 vaccine
3. Fasting Glucose: > 60 - < 125 mg/dl;
4. HbA1C: </= 6.4
5. Vitamin D: > 30 ng/mL
6. Homocysteine < 14 mol/L
7. B12 levels >232 pg/mL
8. Ferritin: > 30 ng/mL
9. Cystatin C: > 0.62 mg/L
10. eGFR > 45 mL/min/1.73 m2
11. BMI > 18 kg/m2 < 35 kg/m²
12. Stable body weight (+/-10 lbs.) over last 6 months
13. Be willing to travel to the study facility as required for this study
14. Be willing to avoid taking antacids 2 hours prior and 2 hours after taking dasatinib
15. Be willing to discontinue proton pump inhibitors
16. Be willing to discontinue St. John's Wort
17. Be willing to discontinue medication/supplements, if applicable, for a washout period and while participating on this study.
18. If taking metformin for anti-aging, willing to washout for 2 months prior to initiating protocol intervention.
19. Be willing to take the investigational product(s) according to schedule and keep a diary for compliance monitoring.
20. Has not participated in another clinical trial within last 30 days
21. If applicable, five years or more post cancer treatment and disease free (define as tumor free or 5 years of clean PET/CT scans).
22. Able to provide signed written informed consent prior to any study specific procedures being performed.

Exclusion Criteria:

1. Inability to provide written informed consent.
2. ECOG score >/= 2
3. More than 1 alcoholic drinks consumed per day.
4. Anemic (defined as hemoglobin (Hb) levels < 12.0 g/dL in women and < 13.0 g/dL in men)
5. Thrombocytopenia (defined as platelet count < 100 × 10^9/L
6. Neutropenia (defined as < 1.0-1.5 × 10^9 neutrophils/L (mild))
7. Any allergy to any medications or supplements used on this trial.
8. Shellfish or iodine allergy (note: glucosamine sulfate supplement contains shellfish (shrimp, crab)
9. Clinically significant vital signs (e.g. uncontrolled hypertension >/= 180/100) or lab abnormalities (defined as platelet count < 100 × 10^9/L; absolute granulocyte count < 1,000/mm3; ALT (SGOT) > 2.0 times the upper limit of normal range; total bilirubin > 2.5 times the upper limit of normal range) at baseline
10. HIV and/or Hepatitis infection
11. Immunosuppressed due to any condition (e.g. transplant).
12. Taking concurrent medications that may interfere with the drugs or supplements used on this study.
13. Any concurrent uncontrolled medical condition or psychiatric illness which could place the patient at unacceptable risk of study treatment.
14. Other concerns that in the PI's judgment will be a potential safety issue for the subject or that precludes the ability to provide informed consent or complete the study.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-06 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events as assessed by CTCAE v5.0 | through study completion, up to post treatment phone (approx. Day 532)
Visceral adipose tissue fat tissue (volume (in^3)) physiological parameter value measured by DEXA scan | Change from baseline to Visit 20 (approx. Day 502)
Systolic blood pressure physiological parameter value measured with a blood pressure cuff | Change from baseline to Visit 20 (approx. Day 502)
Senescent cell-cycle arrest physiological parameter value measured by MMP-9 laboratory test | Change from baseline to Visit 20 (approx. Day 502)
Glucose control (insulin resistance) physiological parameter as measured by HOMA-IR (mg/dL) calculation value | Change from baseline to Visit 20 (approx. Day 502)
  insulin and glucose laboratory values are collected to computer the measurement used
DNA Methylation physiological parameter as measured by 2019 GrimAge Clock laboratory test | Change from baseline to Visit 20 (approx. Day 502)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Anne Weinstock, Study Director — Vitality in Aging

IPD SHARING:
Plan to Share IPD: No